CLINICAL TRIAL: NCT03666494
Title: Ketamine Co-induction for Patients With Major Depressive Disorder; a Randomized Clinical Trial
Brief Title: Ketamine Co-induction for Patients With Major Depressive Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Bio 18-19
Record Dates: First submitted 2018-08-15; First posted 2018-09-11 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Ketamine; Depression; Anesthesia
MeSH Terms: conditions — Depression | interventions — Ketamine; Propofol; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Arm (Active Comparator): As part of the patient's anesthetic induction, they will receive propofol and fentanyl.
  Interventions: Drug: Propofol; Drug: Fentanyl
- Ketamine Arm (Active Comparator): As part of the patient's anesthetic induction, they will receive propofol, fentanyl, as well as ketamine hydrochloride.
  Interventions: Drug: Ketamine Hydrochloride; Drug: Propofol; Drug: Fentanyl

INTERVENTIONS:
Drug: Ketamine Hydrochloride — As part of anesthetic induction, the addition of ketamine hydrochloride 0.5mg/kg.
  Arms: Ketamine Arm
Drug: Propofol — As part of the patient's anesthetic induction, they will receive propofol.
Drug: Fentanyl — As part of the patient's anesthetic induction, they will receive fentanyl.

SUMMARY:
Ketamine hydrochloride, an anesthetic medication, has been demonstrated to acutely and rapidly improve depressive symptoms but not yet been adequately studied for this effect when used as part of a general anesthetic for surgery. This proposed single-centre, double-blinded, randomized clinical trial of adult patients with depression presenting for gynecologic surgery would compare severity of depressive symptoms between patients receiving and not receiving ketamine as part of their general anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder
* Presentation for gynecologic surgery requiring a general anesthetic

Exclusion Criteria:

* Marked co-morbid cardiovascular disease
* Marked co-morbid respiratory disease
* History of intracranial hypertension
* History of seizures
* ASA Physical Status Classification IV or greater
* History of psychosis
* Current pregnancy
* Contraindication to ketamine administration

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Depression Severity | At time of discharge from post-anesthetic care unit, until 3 hours post operatvie
  Severity of depression as measured by Montgomery-Asberg Depression Rating Scale (MADRS), 0-60 where 0 to 6 is normal, 7-19 is mild depression, 20-34 is moderate depression, and >34 is severe depression.
Depression Severity | 72 hours post-operative
  Severity of depression as measured by Montgomery-Asberg Depression Rating Scale (MADRS), 0-60 where 0 to 6 is normal, 7-19 is mild depression, 20-34 is moderate depression, and >34 is severe depression.
Depression Severity | 7-days post-operative
  Severity of depression as measured by Montgomery-Asberg Depression Rating Scale (MADRS), 0-60 where 0 to 6 is normal, 7-19 is mild depression, 20-34 is moderate depression, and >34 is severe depression.
Depression Severity | 30-days post-operative
  Severity of depression as measured by Montgomery-Asberg Depression Rating Scale (MADRS), 0-60 where 0 to 6 is normal, 7-19 is mild depression, 20-34 is moderate depression, and >34 is severe depression.

SECONDARY OUTCOMES:
Pain Score | Pre-operatively
  Verbally reported numeric pain score (out of 10)
Pain Score | Upon discharge from PACU, up to 3 hours postoperative
  Verbally reported numeric pain score (out of 10)
Pain Score | 72 hours post-opertaive
  Verbally reported numeric pain score (out of 10)
Pain Score | 7-days post-op
  Verbally reported numeric pain score (out of 10)
Pain Score | 30-days post-op
  Verbally reported numeric pain score (out of 10)
Analgesia use | Pre-operatively
  Morphine equivalents (in milligrams)
Analgesia use | Upon discharge from PACU, up to 3 hours postoperative
  Morphine equivalents (in milligrams)
Analgesia use | 72 hours post-operative
  Morphine equivalents (in milligrams)
Analgesia use | 7-days post-operative
  Morphine equivalents (in milligrams)
Analgesia use | 30-days post-operative
  Morphine equivalents (in milligrams)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gamble, MD, Principal Investigator — University of Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kudoh A, Takahira Y, Katagai H, Takazawa T. Small-dose ketamine improves the postoperative state of depressed patients. Anesth Analg. 2002 Jul;95(1):114-8, table of contents. doi: 10.1097/00000539-200207000-00020. PMID 12088953
- [Background] McGirr A, Berlim MT, Bond DJ, Fleck MP, Yatham LN, Lam RW. A systematic review and meta-analysis of randomized, double-blind, placebo-controlled trials of ketamine in the rapid treatment of major depressive episodes. Psychol Med. 2015 Mar;45(4):693-704. doi: 10.1017/S0033291714001603. Epub 2014 Jul 10. PMID 25010396
- [Background] Lee EE, Della Selva MP, Liu A, Himelhoch S. Ketamine as a novel treatment for major depressive disorder and bipolar depression: a systematic review and quantitative meta-analysis. Gen Hosp Psychiatry. 2015 Mar-Apr;37(2):178-84. doi: 10.1016/j.genhosppsych.2015.01.003. Epub 2015 Jan 15. PMID 25698228
- [Background] Fond G, Loundou A, Rabu C, Macgregor A, Lancon C, Brittner M, Micoulaud-Franchi JA, Richieri R, Courtet P, Abbar M, Roger M, Leboyer M, Boyer L. Ketamine administration in depressive disorders: a systematic review and meta-analysis. Psychopharmacology (Berl). 2014 Sep;231(18):3663-76. doi: 10.1007/s00213-014-3664-5. Epub 2014 Jul 20. PMID 25038867
- [Background] Larkin GL, Beautrais AL. A preliminary naturalistic study of low-dose ketamine for depression and suicide ideation in the emergency department. Int J Neuropsychopharmacol. 2011 Sep;14(8):1127-31. doi: 10.1017/S1461145711000629. Epub 2011 May 5. PMID 21557878 (Retraction: PMID 28637184 Int J Neuropsychopharmacol. 2017 Jul 1;20(7):611)
- [Background] Caddy C, Giaroli G, White TP, Shergill SS, Tracy DK. Ketamine as the prototype glutamatergic antidepressant: pharmacodynamic actions, and a systematic review and meta-analysis of efficacy. Ther Adv Psychopharmacol. 2014 Apr;4(2):75-99. doi: 10.1177/2045125313507739. PMID 24688759
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270